CLINICAL TRIAL: NCT05815498
Title: A Randomized, Observer-Blind, Active-Controlled Phase 3 Study to Investigate the Safety, Immunogenicity, and Relative Vaccine Efficacy of mRNA-1283 Compared With mRNA-1273 in Participants Aged ≥12 Years for the Prevention of COVID-19
Brief Title: A Study of mRNA-1283 Injection Compared With mRNA-1273 Injection in Participants ≥12 Years of Age to Prevent COVID-19
Acronym: NextCOVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1283-P301; 2023-000884-30 (EudraCT Number)
Record Dates: First submitted 2023-04-13; First posted 2023-04-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: mRNA-1283.222; mRNA-1273.222; mRNA-1283.815; mRNA-1273.815; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: mRNA-1283.222 (Experimental): Participants will receive single intramuscular (IM) injection of mRNA-1283.222 on Day 1.
  Interventions: Biological: mRNA-1283.222
- Part 1: mRNA-1273.222 (Experimental): Participants will receive single IM injection of mRNA-1273.222 on Day 1.
  Interventions: Biological: mRNA-1273.222
- Part 2: mRNA-1283.815 (Experimental): Participants will receive single IM injection of mRNA-1283.815 on Day 1.
  Interventions: Biological: mRNA-1283.815
- Part 2: mRNA-1273.815 (Experimental): Participants will receive single IM injection of mRNA-1273.815 on Day 1.
  Interventions: Biological: mRNA-1273.815

INTERVENTIONS:
Biological: mRNA-1283.222 — Sterile liquid for injection
  Arms: Part 1: mRNA-1283.222
Biological: mRNA-1273.222 — Sterile liquid for injection
  Arms: Part 1: mRNA-1273.222
Biological: mRNA-1283.815 — Sterile liquid for injection
  Arms: Part 2: mRNA-1283.815
Biological: mRNA-1273.815 — Sterile liquid for injection
  Arms: Part 2: mRNA-1273.815

SUMMARY:
The purpose of this study (Part 1 and Part 2) is to evaluate the relative vaccine efficacy (rVE), safety, reactogenicity, and immunogenicity of mRNA-1283.222 versus mRNA-1273.222 (Part 1) and mRNA-1283.815 versus mRNA-1273.815 (Part 2).

ELIGIBILITY:
Key Inclusion Criteria:

* Investigator's assessment that the participant understands and is willing and physically able to comply with protocol-mandated follow-up, including all procedures.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection, and agreement to continue adequate contraception or abstinence through 90 days following the vaccine administration.
* Part 1: Has previously received a primary series of an authorized/approved COVID-19 vaccine. For participants ≥18 years of age, at least 1 booster dose must have also been received. Proof of prior vaccination is required. A heterologous vaccine regimen is acceptable.

Part 2: No prior vaccination is required. For participants who have been previously vaccinated, proof of vaccination is required.

Key Exclusion Criteria:

* Has had close contact, as defined by the Centers for Disease Control and Prevention (CDC), with someone who had a SARS-CoV-2 infection in the past 14 days, or COVID-19 in the past 10 days.
* Participant is acutely ill or febrile (temperature ≥38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
* Any medical, psychiatric, or occupational condition, including reported history of substance abuse, that, in the opinion of the investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 181 days prior to Screening (for corticosteroids ≥10 milligrams (mg)/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Has received or plans to receive any licensed vaccine ≤60 days prior to the study injection (Day 1) or plans to receive a licensed vaccine within 60 days after the study injection.
* Has received systemic immunoglobulins or blood products within 90 days prior to the Screening Visit or plans to receive during the study.
* Has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.
* Has participated in an interventional clinical study within 28 days prior to the Screening Visit based on the medical history interview or plans to do so while participating in this study.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14246 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
Part 1: Geometric Mean Ratio (GMR) of Omicron BA.4/5 mRNA-1283.222 Over the Omicron BA.4/5 mRNA-1273.222 | Day 29
Part 1: Seroresponse Rate (SRR) Difference of Omicron BA.4/5 Between mRNA-1283.222 and mRNA-1273.222 | Day 29
  Seroresponse at the participant level is defined as an antibody value change from baseline below the lower limit of quantification (LLOQ) to ≥4 × LLOQ, or at least a 4-fold rise if baseline is ≥LLOQ and <4 × LLOQ, or at least a 2-fold rise if baseline is ≥4 × LLOQ.
Part 1: GMR of the Ancestral Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) D614G mRNA-1283.222 Over the Ancestral SARS-CoV-2 D614G mRNA-1273.222 | Day 29
Part 1: SRR Difference of Ancestral SARS-CoV-2 D641G Between mRNA-1283.222 and mRNA-1273.222 | Day 29
  Seroresponse at the participant level is defined as an antibody value change from baseline below the LLOQ to ≥4 × LLOQ, or at least a 4-fold rise if baseline is ≥LLOQ and <4 × LLOQ, or at least a 2-fold rise if baseline is ≥4 × LLOQ.
Parts 1 and 2: rVE of mRNA-1283 and mRNA-1273 (Variant Formulations) to Prevent the First Event of COVID-19 | From 14 days after injection to Day 365
  The rVE is defined as the percent of reduction in the hazards of the first occurrence of COVID-19 (mRNA-1283 vs. mRNA-1273) starting 14 days after the booster dose.
Part 1: Number of Participants with Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 7 (7-day follow-up after vaccination)
Part 2: Number of Participants with Solicited Local and Systemic Reactogenicity ARs in Adolescents and Previously Unvaccinated Participants | Up to Day 7 (7-day follow-up after vaccination)
Parts 1 and 2: Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 28 (28-day follow-up after vaccination)
Parts 1 and 2: Number of Participants with Any Serious AEs (SAEs), Medically Attended AEs (MAAEs), AEs Leading to Withdrawal From Study, and AEs of Special Interest (AESIs) | Day 1 to end of study (EOS) (Day 365)

SECONDARY OUTCOMES:
Part 1: Geometric Mean Titers (GMTs) of Omicron BA.4/5 and Ancestral SARS-CoV-2 D614G | Days 91, 181, and 365
Part 1: SRR Against Omicron BA.4/5 and Ancestral SARS-CoV-2 D614G | Days 29, 91, 181, and 365
  Seroresponse at the participant level is defined as an antibody value change from baseline below the LLOQ to ≥4 × LLOQ, or at least a 4-fold rise if baseline is ≥LLOQ and <4 × LLOQ, or at least a 2-fold rise if baseline is ≥4 × LLOQ.
Parts 1 and 2: Number of Participants with a SARS-CoV-2 Infection (Symptomatic or Asymptomatic) | From 14 days after injection to Day 365
Part 2: Number of Participants with Severe COVID-19 | From 14 days after injection to Day 365

CONTACTS AND LOCATIONS:
Locations (229):
- United States (160):
  - Optimal Research, Huntsville, Alabama
  - Accel Research Sites- Achieve Clinical Research, Vestavia Hills, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Phoenix Clinical Research LLC, Phoenix, Arizona
  - FRC - CCT Research, Phoenix, Arizona
  - Headlands Research Sarasota, Scottsdale, Arizona
  - Clinical Research Consortium, Tempe, Arizona
  - Noble Clinical Research, LLC, Tucson, Arizona
  - Del Sol research Management LLC., Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Velocity Clinical Research, Banning, Banning, California
  - Velocity Clinical Research- Chula Vista, Chula Vista, California
  - Benchmark Research, Colton, California
  - Marvel Clinical Research 002, LLC, Huntington Beach, California
  - Velocity Clinical Research Huntington Park, Huntington Park, California
  - Velocity Clinical Research, La Mesa, California
  - Chemidox Clinical Trials, Lancaster, California
  - Long Beach Clinical Trials, Long Beach, California
  - Velocity Clinical Research- Westlake, Los Angeles, California
  - Velocity Clinical Research-North Hollywood, North Hollywood, California
  - Empire Clinical Research, Pomona, California
  - CenExel - CITrials, Riverside, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Benchmark Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Velocity Clinical Research Denver, Denver, Colorado
  - Tekton Research - Fort Collins, Fort Collins, Colorado
  - Tekton Research, Inc- Longmont Center, Longmont, Colorado
  - Alliance for Multispeciality Research - Miami, Coral Gables, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Clinical Research Partners LLC, DeLand, Florida
  - Hillcrest Medical Research, LLC, DeLand, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Sweet Hope Research Specialty, Inc., Hialeah, Florida
  - CenExel Research Centers of America, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Encore Research Group-Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Health Awareness INC, Jupiter, Florida
  - Accel Clinical Research, Lakeland, Florida
  - Accel Research Sites, Largo, Florida
  - Acclaim Clinical Research, Maitland, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Clinical Trials of Florida, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - Clinical Neuroscience Solutions (CNS Healthcare site), Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Pines Care Research Center, Inc., Pembroke Pines, Florida
  - Suncoast Research Associates, LLC, Pembroke Pines, Florida
  - Synexus, Pinellas Park, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Global Health Research Center, Inc., Tampa, Florida
  - Santos Research Center CORP, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Delricht Research, Atlanta, Georgia
  - Atlanta Clinical Research Center, Atlanta, Georgia
  - Baybol Research Institute, Chamblee, Georgia
  - Centricity Research, Columbus, Georgia
  - Elite Research Network, Decatur, Georgia
  - Accel Research Sites Lake Oconee, Eatonton, Georgia
  - Georgia Clinic, PC/CCT Research, Norcross, Georgia
  - Clinical Research Atlanta/Headlands, Stockbridge, Georgia
  - Velocity Clinical Research, Meridian, Idaho
  - Chicago Clinical Research Institute, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Velocity Clinical Research Valparaiso, Valparaiso, Indiana
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - Johnson County Clin-Trials, Inc (JCCT), Lenexa, Kansas
  - Alliance for Multispecialty Research, LLC- Wichita, Wichita, Kansas
  - Tekton Research Inc, Wichita, Kansas
  - Alliance for Multispecialty Research-Lexington, Lexington, Kentucky
  - Versailles Family Medicine, Versailles, Kentucky
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Benchmark Research, Covington, Louisiana
  - MedPharmics, Covington, Louisiana
  - Benchmark Research, Metairie, Louisiana
  - Delricht Research, New Orleans, Louisiana
  - Delricht Clinical Research, Prairieville, Louisiana
  - Centennial Medical Group, Eldridge, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - DM Clinical Research, Brookline, Massachusetts
  - Great Lakes Research Institute, Southfield, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Delricht Research, Gulfport, Mississippi
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Delricht Research, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Delricht Research, Town and Country, Missouri
  - Montana Medical Research, Inc, Missoula, Montana
  - CCT research/ Methodist Physicians Clinic- Prairie Fields, Fremont, Nebraska
  - Velocity Clinical Research, Grand Island, Nebraska
  - Meridian Clinical Research, LLC, Lincoln, Nebraska
  - Velocity Clinical Research, Omaha, Nebraska
  - Papillon Research Centre, Papillion, Nebraska
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - IMA Clinical Research, Warren Township, New Jersey
  - Velocity Clinical Research- New Mexico, Albuquerque, New Mexico
  - IMA Clinical Research, Albuquerque, New Mexico
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - IMA Clinical Research, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research, Inc, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Ohio
  - Tekton Research- Edmond, Edmond, Oklahoma
  - Tekton Research Inc, Moore, Oklahoma
  - Delricht Research, Tulsa, Oklahoma
  - Tekton Research- Yukon, Yukon, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Summit Research Headlands LLC, Portland, Oregon
  - DM Clinical Research, Philadelphia, Pennsylvania
  - Synexus Clinical Research US, Inc, Anderson, South Carolina
  - Velocity Clinical Research-Anderson, Anderson, South Carolina
  - Delricht Research, Charleston, South Carolina
  - Velocity Clinical Research, Columbia, South Carolina
  - Velocity Clinical Research, Greenville, Greenville, South Carolina
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Velocity Clinical Research- Spartanburg, Spartanburg, South Carolina
  - Delricht Research, Hendersonville, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Tekton Research Inc, Austin, Texas
  - Tekton Research - Beaumont, Beaumont, Texas
  - PanAmerican Clinical Research, LLC, Brownsville, Texas
  - Headlands Research Brownsville, Brownsville, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Benchmark Research, Fort Worth, Texas
  - DM Clinical Research, Houston, Texas
  - Ventavia Research Group, Keller, Texas
  - DELRICHT RESEARCH at ZOMNIR FAMILY MEDICINE, McKinney, Texas
  - Research Your Health, Plano, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Tekton Research -San Antonio, San Antonio, Texas
  - DM Clinical Research, Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas
  - Cope Family Medicine, Bountiful, Utah
  - Mountain View Ogden Clinic/CCT Research, Pleasant View, Utah
  - JBR Clinical Research, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Velocity Clinical Research, Portsmouth, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
- Canada (12):
  - Medicor Research Inc., Greater Sudbury, Ontario
  - Hamilton Medical Research group, Hamilton, Ontario
  - Milestone Research Inc., London, Ontario
  - Red Maple Trials Inc., Ottawa, Ontario
  - Winterberry Family Medicine, Stoney Creek, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Centricity Research Toronto Manna Multispecialty, Toronto, Ontario
  - Intermed groupe santé, Chicoutimi, Quebec
  - Centricity Research Pointe-Claire, Pointe-Claire, Quebec
  - Manna Research Inc., Pointe-Claire, Quebec
  - Q&T Research Sherbrooke Inc., Sherbrooke, Quebec
  - Clinique spécialisée en allergie, Québec
- Japan (12):
  - Public Health Association.Inc, Aichi
  - Tenjin Sogo Clinic, Fukuoka
  - Yamasaki Family Clinic - internal medicine, Hyōgo
  - Motomachi Takatsuka Naika Clinic - Internal Medicine, Kanagawa
  - Arakawa Family Clinic, Nagano
  - Koseikai Yotsubashi Clinic - Internal Medicine, Osaka
  - Medical Corporation of Yamazaki Neurotology, Rhinolaryngology Clinic, Sapporo
  - Dojinkinenkai Meiwa Hospital, Tokyo
  - Medical Corporation Asbo Tokyo Asbo Clinic, Tokyo
  - Metropolitan Clinic - Internal Medicine, Tokyo
  - National Center for Global Health and Medicine, Tokyo
  - Shinei Medical Healthcare Clinic, Tokyo
- United Kingdom (45):
  - Barnsley Hospital, Barnsley
  - Royal United Hospital Bath NHS Trust - Royal United Hospital, Bath
  - Layton Medical Centre, Blackpool
  - Dorset Clinical Research Centre (Bournemouth Hospital), Bournemouth
  - Bradford Teaching Hospitals NHS Foundation Trust - Bradford, Bradford
  - Lakeside Healthcare, Corby
  - Rotherham Doncaster and South Humber NHS Foundation Trust, Doncaster
  - University of Dundee - NHS Tayside - Ninewells Hospital & Me, Dundee
  - Western General Hospital, Edinburgh
  - Royal Devon & Exeter Hospital, Exeter
  - CPS Research, Glasgow
  - NHS Greater Glasgow & Clyde, Glasgow
  - Panthera Biopartners - Glasgow - multispeciality, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Gloucestershire Hospitals NHS Foundation Trust - Cheltenham, Gloucester
  - Velocity Clinical Research High Wycombe, High Wycombe
  - University Hospitals of Leicester-Leicester Royal Hospital, Leicester
  - Barts Health NHS Trust, London
  - Egin Research, London
  - Guys and St. Thomas NHS Foundation Trust, London
  - Hammersmith Medicines Research (HMR), London
  - Panthera Biopartners - Enfield, London
  - Richford Gate Medical Practice, London
  - Royal Free London NHS Foundation Trust, London
  - St Georges Healthcare NHS Trust - University of London, London
  - Manchester University NHS Foundation Trust, Manchester
  - Bioluminux Clinical Research, Milton Keynes
  - Stemax Consult Healthcare Services Ltd, Milton Keynes
  - Newcastle University - Institute of Cellular Medicine (ICM), Newcastle
  - Velocity Clinical Research, North London
  - Accellacare North London, Northwood
  - Nottingham University Hospitals NHS Trust - Queens Medical Centre (QMC) Campus, Nottingham
  - Wansford and Kings Cliffe Practice, Peterborough
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Southampton General Hospital - Portsmouth Research Hub, Portsmouth
  - GST NHS Found, Preston
  - Panthera Biopartners Preston, Preston
  - Panthera Biopartners - Manchester - multispeciality, Rochdale
  - Warrington and Halton Teaching hospitals NHS Foundation Trust - Halton General Hospital, Runcorn
  - Panthera Biopartners - Sheffield - multispeciality, Sheffield
  - Royal Victoria Infirmary, Sheffield
  - Southampton University Hospital NHS Foundation Trust, Southampton
  - Pier Health Group, Weston-super-Mare
  - Weymouth Research Hub, Weymouth
  - North Wales Clinical Research Centre, Wrexham

REFERENCES:
- [Derived] Chalkias S, Dennis P, Petersen D, Radhakrishnan K, Vaughan L, Handforth R, Rossi A, Wahid R, Edwards DK, Feng J, Deng W, Zhou H, De Windt E, Urdaneta V, Paila Y, Girard B, Faust SN, Walsh SR, Cosgrove CA, Miller J, Das R. Efficacy, immunogenicity, and safety of a next-generation mRNA-1283 COVID-19 vaccine compared with the mRNA-1273 vaccine (NextCOVE): results from a phase 3, randomised, observer-blind, active-controlled trial. Lancet Infect Dis. 2025 Nov;25(11):1230-1242. doi: 10.1016/S1473-3099(25)00236-1. Epub 2025 Jul 7. PMID 40639387